CLINICAL TRIAL: NCT01227941
Title: A Phase Ib Dose Escalation Study of MK-4827 in Combination With Pegylated Liposomal Doxorubicin (Doxil™ or Caelyx™) in Patients With Advanced Solid Tumors With a Cohort Expansion in Patients With Platinum Resistant/Refractory High Grade Serous Ovarian Cancer
Brief Title: MK-4827 in Combination With Pegylated Liposomal Doxorubicin in Participants With Advanced Solid Tumors and Ovarian Cancer (MK-4827-011)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-4827-011
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2012-03

CONDITIONS: Ovarian Cancer
Keywords: advanced solid tumors; ovarian cancer; pegylated liposomal doxorubicin; Doxil; Caelyx
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: MK-4827 + pegylated liposomal doxorubicin (Experimental): MK-4827 and pegylated liposomal doxorubicin combination. Dose escalation/confirmation in participants with advanced solid tumors
  Interventions: Drug: MK-4827 + pegylated liposomal doxorubicin
- Part B: MK-4827 + pegylated liposomal doxorubicin (Experimental): MK-4827 and pegylated liposomal doxorubicin combination at 1 or 2 dose levels of MK-4827 to be determined from the results of Part A. Ovarian Cancer Cohort
  Interventions: Drug: MK-4827 + pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: MK-4827 + pegylated liposomal doxorubicin — Initial evaluation of a 16-day dosing schedule: A loading dose of MK-4827 will be administered orally on Days 1-2 of the cycle and a maintenance dose daily on Days 3-16. Pegylated liposomal doxorubicin 40 mg/m^2 will be administered intravenously on Day 3 of each cycle. The maintenance dose of MK-4827 will be escalated, until the maximum tolerated dose (MTD) is determined. If the maintenance dose is escalated above the loading dose, the loading dose will be escalated to a level equal to the maintenance dose, for the subsequent cycle. Other dosing schedules of MK-4827 may be explored, including 7-, 10-, 21- and 28-day schedules.
  Other Names: Doxil, Caelyx
  Arms: Part A: MK-4827 + pegylated liposomal doxorubicin
Drug: MK-4827 + pegylated liposomal doxorubicin — MK-4827 will be administered according to one or two dose schedules as determined in Part A. Pegylated liposomal doxorubicin 40 mg/m^2 will be administered intravenously on Day 3 of the cycle.
  Other Names: Doxil, Caelyx
  Arms: Part B: MK-4827 + pegylated liposomal doxorubicin

SUMMARY:
This study will determine whether MK-4827 can be safely administered in combination with pegylated liposomal doxorubicin, and if so, will obtain an estimate of the benefit of the combination in patients with ovarian cancer as compared to historical data with single agent pegylated liposomal doxorubicin. The first part of the study (Part A) is designed to determine the maximum tolerated dose (MTD) and evaluate the safety of MK-4827, when administered in combination with pegylated liposomal doxorubicin. Part B is designed to assess preliminary clinical activity of MK-4827, when administered in combination with pegylated liposomal doxorubicin to participants with ovarian cancer. It is hypothesized that MK-4827 can be administered, in conjunction with pegylated liposomal doxorubicin, with acceptable tolerability and that MK-4827, administered in conjunction with pegylated liposomal doxorubicin, will demonstrate a tumor response rate equal or superior to that of historical data for pegylated liposomal doxorubicin alone.

DETAILED DESCRIPTION:
The decision to discontinue new enrollment is not related to any concerns about the safety profile of the product.

ELIGIBILITY:
Inclusion Criteria:

Parts A and B:

* The participant has a locally advanced or metastatic solid tumor and lacks curative options

  * Pegylated liposomal doxorubicin must be an appropriate therapy or the participant has not responded to standard of care or therapies known to provide clinical benefit, or has refused such therapies or no therapy is known to provide clinical benefit
* Part B only: Female participants must have high grade serous ovarian cancer without curative options; pegylated liposomal doxorubicin must be an appropriate therapy. Eligible patients for Part B must have:

  * Platinum-resistant ovarian cancer, defined as tumor progression within 6 months of completing treatment with a platinum-containing agent, OR secondary platinum-refractory ovarian cancer defined as tumor progression while on treatment for recurrent ovarian cancer after initially responding to a platinum-based chemotherapy regimen in the first line setting; and
  * Measurable disease, OR elevated serum cancer antigen 125 (CA-125) levels at baseline, defined as a pre-treatment sample that is at least twice the upper limit of normal and within 2 weeks prior to starting treatment
  * Participant has a performance status of 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) Performance Scale
  * Participant must have adequate organ function
  * Participant has no history of a prior malignancy with the exception of cervical intraepithelial neoplasia, basal cell carcinoma of the skin, or has undergone potentially curative therapy with no evidence of that disease for five years, or is deemed at low risk for recurrence by his/her treating physician

Exclusion Criteria:

Parts A and B:

The participant:

* Has had chemotherapy, radiotherapy, or biological therapy within 4 weeks of entering the study
* Has previously been treated with pegylated liposomal doxorubicin
* Has active central nervous system metastases or a primary central nervous system tumor
* Part A: Has had more than two prior chemotherapy regimens; in Part B, there is no limit to the number of prior chemotherapy regimens
* Is known to be Human Immunodeficiency Virus (HIV) positive
* Has a known history of Hepatitis B or C
* Has a left ventricular ejection fraction (LVEF) below the institutional lower limit of normal
* Has had prior doxorubicin exposure >240 mg/m^2 (or anthracycline equivalent)
* Has initiated or adjusted bisphosphonate therapy/regimen within 30 days prior to Cycle 1 Day 1
* Part B only: Has been previously treated with a poly[ADP] ribose polymerase (PARP) inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) | 28 days (one cycle of treatment)
Tumor response rate | Every 8 weeks until disease progression
  A tumor response is defined as a complete response, partial response, or a sustained decrease in tumor marker levels.